CLINICAL TRIAL: NCT03951350
Title: Effectiveness and Cost-effectiveness of a Lifestyle Modification Program in the Prevention and Treatment of Subclinical, Mild and Moderate Depression in Primary Care: A Randomized Clinical Trial Protocol
Brief Title: Lifestyle Modification Program in the Prevention and Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Bárbara Oliván-Blázquez, Professor University of Zaragoza, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI18/01336
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Lifestyle modifications; Depression; primary health care; Diet; Exercise; Sunlight exposure; Sleep patterns
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (TAU) (No Intervention): Patients will follow the usual treatment provided by their GP (treatment-as-usual, TAU).
- Lifestyle Modification Program (LMP) (Experimental): It will consist of 6 weekly group sessions (lasting 90 minutes each).
  Interventions: Behavioral: Lifestyle Modification Program (LMP); Behavioral: Lifestyle Modification Program (LMP) + Information Communication Technologies (ICTs)
- Lifestyle Modification Program (LMP) + ICTs (Experimental): It will consist of 6 weekly group sessions (lasting 90 minutes each).
  Interventions: Behavioral: Lifestyle Modification Program (LMP) + Information Communication Technologies (ICTs)

INTERVENTIONS:
Behavioral: Lifestyle Modification Program (LMP) — Patients will follow TAU and LMP. This program will consist of 6 weekly group sessions (lasting 90 minutes each) led by an experienced psychologist and complemented by PowerPoint presentations. The content is the following:
  1. Presentation of the project and psychoeducation on depression.
  2. Behavior activation.
  3. Sleep hygiene habits and careful exposure to sunlight.
  4. Physical activity.
  5. Adherence to the Mediterranean diet.
  6. Summary of previous sessions with practical final suggestions.
  Arms: Lifestyle Modification Program (LMP)
Behavioral: Lifestyle Modification Program (LMP) + Information Communication Technologies (ICTs) — Patients will follow TAU and LMP and will be monitored using a wearable smart wristwatch that will track their daily sleep patterns and physical activity (LMP+ICTs).
  Arms: Lifestyle Modification Program (LMP); Lifestyle Modification Program (LMP) + ICTs

SUMMARY:
Introduction:

Major depression is a highly prevalent pathology that is currently the second most common cause of disease-induced disability in our society. The onset and continuation of depression may be related to a wide variety of biological and psychosocial factors, many of which are linked to different lifestyle aspects. Therefore, health systems must design and implement health promotion and lifestyle modification programs, taking into account personal factors and facilitators. The main objective of this work is to analyze the utility and cost-effectiveness of an adjunctive treatment program for subclinical, mild or moderate depression in Primary Care patients, based on healthier lifestyle recommendations. Secondary objectives include the analysis of the effectiveness of the intervention in comorbid chronic pathology and the measurement of the influence of personal factors on lifestyle modification.

Methods and analysis:

A randomized, multicenter pragmatic clinical trial with 3 parallel groups consisting of primary healthcare patients suffering from subclinical, mild or moderate depression. The following interventions will be used: 1. Usual antidepressant treatment with psychological advice and/or psychotropic drugs prescribed by the General Practitioner (treatment-as-usual, TAU). 2. TAU + Lifestyle Modification Program (LMP). A program to be imparted in 6 weekly 90-minute group sessions, intended to improve the following aspects: behavioral activation + daily physical activity + adherence to the Mediterranean diet pattern + sleep hygiene + careful exposure to sunlight. 3. TAU + LMP + ICTs: healthy lifestyle recommendations (TAU+LMP intervention) + monitoring using ICTs (a wearable smartwatch). The primary outcome will be the depressive symptomatology and the secondary outcomes will be the quality of life, the use of health and social resources, personal variables related to program adherence (patient activation in their own health, self-efficacy, sense of coherence, health literacy and procrastination) and chronic comorbid pathology. Data will be collected before and after the intervention, with 6- and 12-month follow-ups.

ELIGIBILITY:
Inclusion criteria:

* Individuals over the age of 18.
* Both sexes.
* Having a duration of depression symptoms of at least 2 months.
* Who perfectly understand written and spoken Spanish.
* Who have provided their informed consent.

Exclusion criteria:

* Suffering from another disease that affects the central nervous system (organic brain pathology or having suffered a traumatic brain injury of any severity, dementia).
* Having another psychiatric diagnosis or serious psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders) with the exception of anxious pathology or personality disorders (collected through a medical history and from the Mini-International Neuropsychiatric Interview (MINI) (Ferrando, Bobes, & Gibert, 2000)).
* Presence of a serious or uncontrolled medical, infectious or degenerative illness that may interfere with the affective symptoms.
* Presence of delirium or hallucinations, risk of suicide, pregnancy or lactation.
* Patients who have participated in another clinical trial over the past 6 months or who are currently in psychotherapy.
* Who practice mindfulness, yoga, meditation or similar practices over the past 6 months, engaging in formal practice at least once a week.
* Presence of any medical, psychological or social problem that could seriously interfere with the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Beck II Self-Applied Depression Inventory (BDI-II) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  The primary outcome will be measured using the BDI-II (Beck et al., 1996). This is a self-report inventory for measuring the severity of depression, consisting of 21 multiple-choice questions with each answer being scored on a scale ranged from 0 to 3. It was translated and validated into Spanish with a reliability of .89 (Sanz et al., 2005). The standardized cutoffs are: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.

SECONDARY OUTCOMES:
International Neuropsychiatric Interview (MINI) | Baseline
  It is a short-term structured diagnostic interview that explores the main psychiatric disorders of Axis I of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and International Classification of Diseases (ICD-10) (Ferrando et al., 2000).
Comorbidity with chronic diseases | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Comorbidity with chronic diseases will be determined according to the International Classification of Diseases (ICD-10) (WHO, 2010): diabetes (glucose concentration (mg/dl), glycated hemoglobin (%), creatinine), arterial hypertension and diseases of lipid metabolism. In patients with chronic heart disease, coagulation variables will be added. They will be collected from the last blood test or control measurements of the clinical history, taken by their general practitioner (GP) or nurse (assuming they were taken over the past 3 months). Otherwise, their GP will be asked for a blood control test. It is estimated that approximately 50% of these patients will present some comorbidity (Katon, 2003). Anthropometric measures will also be collected (weight, size and perimeter of the waist).
European Quality of Life-5 Dimensions questionnaire (EQ-5D) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Health-related quality of life will be measured using the European Quality of Life-5 Dimensions questionnaire (EQ-5D) (Brooks & De Charro, 1996; The EuroQol Group, 1990). EQ-5D scores will be used to calculate the quality-adjusted life year (QALY) during the monitoring period by adjusting the length of time affected by the health result by the utility value. It contains five health dimensions (mobility, selfcare, usual activities, pain/discomfort and anxiety/depression) and each of these has three levels (no problems, slight problems or moderate and severe problems). The EQ records the patient's self-rated health on a vertical visual analogue scale of 20 centimeters (VAS). The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgment. Patients mark the point on the vertical line that best reflects their assessment of their current global health status (Badia, Roset, Montserrat, Herdman, & Segura, 1999).
Physical activity questionnaire (IPAQ-SF) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Physical activity will be measured using the International Physical Activity Questionnaire-Short Form (IPAQ-SF) (Kim, Park, & Kang, 2013). It assesses the levels of habitual physical activity over the last 7 days. It has 7 items and records the activity of four intensity levels: vigorous-intensity activity, moderate-intensity activity (walking and sitting). We will use the validated Spanish version (Roman-Viñas et al., 2010). IPAQ-SF has acceptable validity for the measurement of total and vigorous physical activity and poor validity for moderate activity and good reliability (Kurtze, Rangul, & Hustvedt, 2008).
Mediterranean Diet Adherence Screener (MEDAS) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using the 14-item Mediterranean Diet Adherence Screener (MEDAS), developed within the PREDIMED study group (Martínez-González et al., 2010). It includes items on food consumption and intake habits: the use of olive oil as the main source of cooking fat, preference for white meat over red meat, servings of vegetables, portions of fruit, red meat or sausages, servings of animal fat, sugar-sweetened beverages, red wine, legumes, fish, commercial pastries and dressing food with a traditional sauce made of tomatoes, garlic, onion, or leeks sautéed in olive oil. The total score ranges from 0 to 14, with a higher score indicating a better accordance with the Mediterranean diet (Schröder et al., 2011).
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using the Pittsburgh Sleep Quality Index (PSQI) (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). To measure sleep quality and patterns in adults. It differentiates between "poor" and "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the past month. It consists of 19 self-applied questions and 5 questions that request the evaluation of the patient's bedmate or roommate (these are not scored). Answers range from 0 (no difficulty) to 3 (severe difficulty). The overall score ranges from 0 to 21 points. In its Spanish version, the Cronbach's alpha coefficient is .81, sensitivity of 88.63% and specificity of 74.99%. We will use the validated Spanish version (Royuela Rico & Macías Fernández, 1997).
Patient Activation Questionnaire (PAM) in relation to the management of their health | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using the Patient Activation Questionnaire (PAM) with regard to the management of their health. It evaluates the patient's perceived knowledge, skills, and confidence to engage in self-management activities. It has 13 items, a Likert scale from 1 (strongly disagree) to 4 (strongly agree). The resulting score (between 0 and 100) places the individual at one of four levels of activation, each of which reveals insight into a range of health-related characteristics, including behaviors and outcomes. Higher scores indicate higher levels of activation (Hibbard et al., 2004). This scale is only validated in Spanish for chronic patients. It had an item separation index for the parameters of 6.64 and a reliability of .98 (Moreno Chico, González de Paz, Monforte Royo, Navarro Rubio, & Gallart Fernández Puebla, 2018).
Social support questionnaire (MOS) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  It will be measured by the Medical Outcomes Study Social Support Survey (MOS-SS) (Sherbourne & Stewart, 1991). It is a self-report instrument consisting of four subscales (emotional/informational, tangible, affectionate, and positive social interaction) and an overall functional social support index. It has a good reliability (Cronbach's alpha ≥ .91) and is quite stable over time. It has 19 items, a five-point Likert scale. Higher scores indicate more support. We will use the Spanish validated version (de la Revilla-Ahumada L, Luna del Castillo J, & Bailón Muñoz E, 2005).
The Self-Efficacy Scale | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using by the Self-Efficacy Scale (Sherer et al., 1982). To measure General Self-Efficacy subscale (17 items including individuals' beliefs in their ability to perform well in a variety of situations) and Social Self-Efficacy subscale (6 items). It contains 23 items that are rated on a 14-point scale (ranging from strongly agree to strongly disagree). Higher scores indicate higher levels of self-efficacy. It has a Cronbach coefficient alpha of .86 for General Self-efficacy subscale and .71 for the Social Self-efficacy subscale. The unpublished Spanish version was translated by Godoy in 1990 (Lopez-Torrecillas, García, Cañadas, Ramirez Ucles, & de la Fuente, 2006).
Sense of coherence questionnaire of Antonovsky | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using the Sense of Coherence (SOC) questionnaire by Antonovsky (Antonovsky, 1993). It values the personal disposition towards the assessment of vital experiences. It measures the sense of coherence, comprehensibility, manageability and meaningfulness. It has 13 items scoring between 13 and 91 points. It has consistency rates of between .84 and .93. Higher scores (after reversal of the inverted items) indicate a higher sense of coherence. We will use the validated Spanish version (Moreno, B., Alonso, M., & Álvaréz, 1997).
Health Literacy Europe questionnaire (HLS-EUQ16) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using the Health Literacy Europe Questionnaire (HLS-EUQ16) (Sørensen et al., 2015). It can indicate that the probability of functional literacy in limited health is high, a possibility of functional literacy in limited health, and a functional health literacy in adequate health. It contains 16 items. Higher scores indicate better health literacy. It presents a high consistency (Cronbach's alpha of .982) in the Spanish validation (Nolasco et al., 2018).
Irrational Procrastination Scale (IPS) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  Measured using the Irrational Procrastination Scale (IPS) (Steel, 2010). To measure general procrastination (dysfunctional delay). It has 9 items, rated on a 5-point Likert scale, with higher scores (after reversal of the three procrastination-inconsistent items) indicating a higher level of procrastination. Its Cronbach's alpha value is 0.90. We will use the validated Spanish version (Guilera et al., 2018).
Client Service Receipt Inventory (CSRI) | Change from baseline, immediately after the intervention and at six and 12-month follow-up.
  It will be measured using the Client Service Receipt Inventory (CSRI) (Knapp, 2001). This data may be used for a wide range of applications, including estimates of the costs of service receipt. To collect information on the entire range of services and supports used by study participants. It retrospectively collects data on the use of services over the past 6 months (e.g., rates of use of individual services, mean intensity of service use, rates of accommodation use over time). We will use the validated Spanish version (Vazquez-Barquero, Gaite, Cuesta, Garcia, & Knapp, 1997).

CONTACTS AND LOCATIONS:
Locations (1):
- Alejandra Aguilar-Latorre, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Proposals should be directed to barbaraolivan@gmail.com. To gain access, data requestors will need to sing a data access agreement. Data will be available for 5 years after we publish the results.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Sanz J, Garcia Vera MP, Espinosa R, Fortun M, Vazquez C. Adaptación española del Inventario para la Depresión de Beck II: Propiedades psicométricas en pacientes con trastornos psicológicos. Clínica y Salud 2005; 16: 121-42.
- [Background] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Background] Drummond MF, Sculpher MJ, Torrance GW, O'Brien B, Stoddart GL: Methods for the Economic Evaluation of Health Care Programmes. Oxford, Oxford University Press; 2005.
- [Background] Kim Y, Park I, Kang M. Convergent validity of the international physical activity questionnaire (IPAQ): meta-analysis. Public Health Nutr. 2013 Mar;16(3):440-52. doi: 10.1017/S1368980012002996. Epub 2012 Jul 2. PMID 22874087
- [Background] Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ros E, Covas MI, Fiol M, Warnberg J, Aros F, Ruiz-Gutierrez V, Lamuela-Raventos RM, Lapetra J, Munoz MA, Martinez JA, Saez G, Serra-Majem L, Pinto X, Mitjavila MT, Tur JA, Portillo MP, Estruch R; PREDIMED Study Investigators. Cohort profile: design and methods of the PREDIMED study. Int J Epidemiol. 2012 Apr;41(2):377-85. doi: 10.1093/ije/dyq250. Epub 2010 Dec 20. No abstract available. PMID 21172932
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Sherer M, Maddux JE, Mercandante B, Prentice-Dunn S, Jacobs B, Rogers RW. The Self-Efficacy Scale: Construction and Validation. Psychol Rep 1982;51(2):663 -71.
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Antonovsky A. The structure and properties of the sense of coherence scale. Soc Sci Med. 1993 Mar;36(6):725-33. doi: 10.1016/0277-9536(93)90033-z. PMID 8480217
- [Background] Sorensen K, Pelikan JM, Rothlin F, Ganahl K, Slonska Z, Doyle G, Fullam J, Kondilis B, Agrafiotis D, Uiters E, Falcon M, Mensing M, Tchamov K, van den Broucke S, Brand H; HLS-EU Consortium. Health literacy in Europe: comparative results of the European health literacy survey (HLS-EU). Eur J Public Health. 2015 Dec;25(6):1053-8. doi: 10.1093/eurpub/ckv043. Epub 2015 Apr 5. PMID 25843827
- [Background] Guilera G, Barrios M, Penelo E, Morin C, Steel P, Gomez-Benito J. Validation of the Spanish version of the Irrational Procrastination Scale (IPS). PLoS One. 2018 Jan 5;13(1):e0190806. doi: 10.1371/journal.pone.0190806. eCollection 2018. PMID 29304119
- [Background] Ferrando, L., Bobes, J., Gibert, J., Soto, M. y Soto, O. (2000). MINI. Entrevista Neuropsiquiátrica Internacional. Versión en Español 5.0.0. DSM-IV. Traducida por L. Franco-Alfonso, L. Franco. Bajada de http://entomologia.rediris.es /pub/bscw.cgi/ d602335/ MINI/Entrevista Neuropsiquiátrica Internacional.pdf
- [Background] WHO. (2010). International Classification of Diseases (ICD-10). Family Practice Management.
- [Background] Katon WJ. Clinical and health services relationships between major depression, depressive symptoms, and general medical illness. Biol Psychiatry. 2003 Aug 1;54(3):216-26. doi: 10.1016/s0006-3223(03)00273-7. PMID 12893098
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Roman-Viñas, B., Serra-Majem, L., Hagströmer, M., Ribas-Barba, L., Sjöström, M., & Segura-Cardona, R. (2010). International physical activity questionnaire: Reliability and validity in a Spanish population. European Journal of Sport Science, 10(5), 297-304. https://doi.org/10.1080/17461390903426667
- [Background] Kurtze N, Rangul V, Hustvedt BE. Reliability and validity of the international physical activity questionnaire in the Nord-Trondelag health study (HUNT) population of men. BMC Med Res Methodol. 2008 Oct 9;8:63. doi: 10.1186/1471-2288-8-63. PMID 18844976
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Knapp, M. (2001). Economic Evaluation of Mental Health Care. In Contemporary Psychiatry. https://doi.org/10.1007/978-3-642-59519-6_16
- [Background] de la Revilla-Ahumada L, Luna del Castillo J, Bailón Muñoz E, M. M. I. (2005). [Validation of a questionnaire to measured social support in Primary Care]. Medicina de Familia (Andalucía).
- [Background] Royuela Rico, A., & Macías Fernández, J. A. (1997). Propiedades clinimétricas de la versión castellana del Cuestionario de Pittsburgh. Vigilia-Sueño.
- [Background] Moreno Chico, C., González de Paz, L., Monforte Royo, C., Navarro Rubio, M. D., & Gallart Fernández Puebla, A. (2018). Adaptación y validación de la escala de evaluación de la activación "Patient Activation Measure 13" (PAM13) en una muestra de pacientes crónicos visitados en CAP Rambla de MútuaTerrassa. XXIV Premi d'infermeria 2018.
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Lopez-Torrecillas F, Garcia J, Canadas GA, Ucles IR, De La Fuente EI. Validity of self-efficacy scale scores for a Spanish sample. Psychol Rep. 2006 Apr;98(2):437-50. doi: 10.2466/pr0.98.2.437-450. PMID 16796100
- [Background] Moreno, B., Alonso, M., & Álvaréz, E. (1997). Sentido de coherencia, personalidad resistente, autoestima y salud. Revista de Psicología de La Salud, 9(2), 115-137.
- [Background] Nolasco A, Barona C, Tamayo-Fonseca N, Irles MA, Mas R, Tuells J, Pereyra-Zamora P. [Health literacy: psychometric behaviour of the HLS-EU-Q16 questionnaire]. Gac Sanit. 2020 Jul-Aug;34(4):399-402. doi: 10.1016/j.gaceta.2018.08.006. Epub 2018 Nov 22. Spanish. PMID 30473252
- [Background] Steel, P. (2010). Arousal, avoidant and decisional procrastinators: Do they exist? Personality and Individual Differences. https://doi.org/10.1016/j.paid.2010.02.025
- [Background] Vazquez-Barquero, J. L., Gaite, L., Cuesta, M. J., Garcia, U. E., & Knapp, M. (1997). Spanish version of the CSRI: A mental health cost evaluation interview. [Spanish version of the CSRI: A mental health cost evaluation interview.]. Archivos de Neurobiología.
- [Derived] Aguilar-Latorre A, Olivan-Blazquez B, Algorta GP, Serrano-Ripoll MJ, Olszewski LE, Turon-Lanuza A. One-year follow-up of the effectiveness of a lifestyle modification programme as an adjuvant treatment of depression in primary care: A randomised clinical trial. J Affect Disord. 2023 Jul 1;332:231-237. doi: 10.1016/j.jad.2023.04.007. Epub 2023 Apr 11. PMID 37054898
- [Derived] Aguilar-Latorre A, Navarro C, Olivan-Blazquez B, Gervilla E, Magallon Botaya R, Calafat-Villalonga C, Garcia-Toro M, Boira S, Serrano-Ripoll MJ. Effectiveness and cost-effectiveness of a lifestyle modification programme in the prevention and treatment of subclinical, mild and moderate depression in primary care: a randomised clinical trial protocol. BMJ Open. 2020 Dec 28;10(12):e038457. doi: 10.1136/bmjopen-2020-038457. PMID 33372070